CLINICAL TRIAL: NCT03841981
Title: Amount, Distribution and Dysfunction of Body Fat as Determinants of Female Gonadal Dysfunction: From Functional Hypothalamic Amenorrhea to the Polycystic Ovary Syndrome
Brief Title: Body Fat as Determinant of Female Gonadal Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); University of Alcala (Other)
Responsible Party: Sponsor
Other Study IDs: PI18/01122
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome; Hypothalamic Amenorrhea
Keywords: Exercise; Sex steroids; Hyperandrogenism; Adipose tissue; Muscle; Proteome; Gene expression; Adipokine; Cardiovascular risk; Microbiome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity; Hyperandrogenism | interventions — Physical Examination; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Plasma Whole blood samples Subcutaneous adipose tissue by percutaneous biopsy Muscle tissue by percutaneous biopsy Feces Oral smear
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- I- Hypothalamic amenorrhea: 10 women with exercise-associated hypothalamic amenorrhea
  Interventions: Diagnostic Test: Anthropometric and physical examination; Diagnostic Test: Indirect calorimetry, accelerometer and seven-day dietary recall; Diagnostic Test: Biochemical, hormonal and metabolic phenotyping; Diagnostic Test: Sonographic studies; Diagnostic Test: 24-hour Ambulatory blood pressure monitoring; Procedure: Percutaneous biopsy; Diagnostic Test: Cardiovascular autonomic function studies; Diagnostic Test: Oral smear and feces specimen
- II- Hyperandrogenic polycystic ovary syndrome: 5 lean women with hyperandrogenic polycystic ovary syndrome. 5 women with weight excess and hyperandrogenic polycystic ovary syndrome.
  Interventions: Diagnostic Test: Anthropometric and physical examination; Diagnostic Test: Indirect calorimetry, accelerometer and seven-day dietary recall; Diagnostic Test: Biochemical, hormonal and metabolic phenotyping; Diagnostic Test: Sonographic studies; Diagnostic Test: 24-hour Ambulatory blood pressure monitoring; Procedure: Percutaneous biopsy; Diagnostic Test: Cardiovascular autonomic function studies; Diagnostic Test: Oral smear and feces specimen
- III- Non-hyperandrogenic polycystic ovary syndrome: 5 lean women with non-hyperandrogenic polycystic ovary syndrome 5 women with weight excess and non-hyperandrogenic polycystic ovary syndrome
  Interventions: Diagnostic Test: Anthropometric and physical examination; Diagnostic Test: Indirect calorimetry, accelerometer and seven-day dietary recall; Diagnostic Test: Biochemical, hormonal and metabolic phenotyping; Diagnostic Test: Sonographic studies; Diagnostic Test: 24-hour Ambulatory blood pressure monitoring; Procedure: Percutaneous biopsy; Diagnostic Test: Cardiovascular autonomic function studies; Diagnostic Test: Oral smear and feces specimen
- IV- Trained women without ovulatory dysfunction: 10 women who exercise as intensively as women with exercise-associated hypothalamic amenorrhea but with normal ovulatory cycles.
  Interventions: Diagnostic Test: Anthropometric and physical examination; Diagnostic Test: Indirect calorimetry, accelerometer and seven-day dietary recall; Diagnostic Test: Biochemical, hormonal and metabolic phenotyping; Diagnostic Test: Sonographic studies; Diagnostic Test: 24-hour Ambulatory blood pressure monitoring; Procedure: Percutaneous biopsy; Diagnostic Test: Cardiovascular autonomic function studies; Diagnostic Test: Oral smear and feces specimen
- V- Non-hyperandrogenic healthy women: 10 women matched by age and body mass index with women with polycystic ovary syndrome who do not perform physical activity on a regular basis
  Interventions: Diagnostic Test: Anthropometric and physical examination; Diagnostic Test: Indirect calorimetry, accelerometer and seven-day dietary recall; Diagnostic Test: Biochemical, hormonal and metabolic phenotyping; Diagnostic Test: Sonographic studies; Diagnostic Test: 24-hour Ambulatory blood pressure monitoring; Procedure: Percutaneous biopsy; Diagnostic Test: Cardiovascular autonomic function studies; Diagnostic Test: Oral smear and feces specimen

INTERVENTIONS:
Diagnostic Test: Anthropometric and physical examination — * Weight and height.
  * Waist-to-hip ratio.
  * Body composition: Bioelectrical impedance and [Dual energy X-ray absorptiometry (DEXA)].
Diagnostic Test: Indirect calorimetry, accelerometer and seven-day dietary recall — Energy availability assessment.
Diagnostic Test: Biochemical, hormonal and metabolic phenotyping — * Lipid profile.
  * Oral glucose tolerance test: plasma glucose and insulin, insulin sensitivity indices, gastrointestinal hormones, adipokines, oxidative stress markers.
  * Sex steroid profile.
  * Hypothalamic-pituitary-adrenal axis study.
  * Ferrokinetic study.
  * Subclinical chronic inflammatory markers.
Diagnostic Test: Sonographic studies — * Polycystic ovarian morphology.
  * Carotid intima-media thickness.
  * Eco-FAT: Ultrasound measurements of adipose tissue depots including sc, preperitoneal, intraperitoneal (ip), mesenteric, and perirenal fat thickness.
Diagnostic Test: 24-hour Ambulatory blood pressure monitoring — A&D TM2430EX oscillometric devices (A&D Company Limited, Tokyo, Japan).
Procedure: Percutaneous biopsy — Subcutaneous fat tissue and muscle tissue for proteomics an gene expression studies.
Diagnostic Test: Cardiovascular autonomic function studies — Parasympathetic and sympathetic responses to deep breathing, Valsalva's maneuver and orthostatism.
Diagnostic Test: Oral smear and feces specimen — Microbiome studies.

SUMMARY:
Reproduction requires from women enough energy depots to warrant an adequate nutritional supply to the fetus. Hence, adipose tissue is able to communicate with female hypothalamic-pituitary-ovary axis. The hypothesis of the project is that abnormalities in the quantity (absolute and relative to lean body mass), distribution and/or function of adipose tissue are associated with functional forms of female gonadal dysfunction in predisposed women, in a spectrum of anomalies that go from hypothalamic amenorrhea to the polycystic ovary syndrome (PCOS). To challenge this hypothesis, the investigators will study 5 groups of 10 women each: women with exercise-associated hypothalamic amenorrhea, women without ovulatory dysfunction that exercise equally, non-hyperandrogenic patients with PCOS, hyperandrogenic patients with PCOS, and healthy control women comparable to those with PCOS. The aims of the study will be:

Primary objective: To identify novel signalling factors originating from adipose tissue and muscle using targeted and nontargeted evaluation of the proteome and of gene expression of superficial subcutaneous fat, deep subcutaneous fat (which mimics visceral adipose tissue) and skeletal muscle.

Secondary objectives:

1. To study the serum adipokine profile - including those identified by the primary objective - and circulating gut hormones during fasting and after a glucose load in the 5 groups of women, and their associations with sexual hormones and body fat distribution.
2. To study body composition and body fat distribution in these women and their relationships with:

2.1, Sex steroid profiles.

2.2. Classic cardiovascular risk factors: carbohydrate metabolism, lipid profiles and blood pressure.

2.3 Markers of low-grade chronic inflammation.

2.4. Oxidative stress markers.

2.5. Cardiovascular autonomic function.

2.6. Surrogate markers of subclinical atherosclerosis.

2.7. Circulating concentrations of endocrine disruptors.

2.8. Oral and gut microbiome.

The results will provide a better understanding of the mechanisms linking body energy depots with the female reproductive axis and, hopefully, the identification of potential biomarkers for the diagnosis and treatment of the disorders studied here.

ELIGIBILITY:
Inclusion Criteria

Group I

* Body mass index between 18.5 and 25.0 kg/m2.
* Group 1 ovulatory dysfunction [World Health Organization (WHO) classification].
* Normal/low gonadotrophin levels [follicle-stimulating hormone (FSH) and luteinizing (LH) < 10 IU/l] and low estradiol (< 50 pg/ml).
* Moderate-vigorous intensity physical activity (> 5 hours per week) plus low energy availability (< 30 kcal/per kg of lean mass).
* Exclusion of secondary etiologies
* Informed consent signed.

Group II:

* Polycystic ovary syndrome phenotype I, II and III [National Institute of Health (NIH)-2012] with hyperandrogenemia (http://prevention.nih.gov/workshops/2012/resources.aspx).
* Body mass index between 18.5 and 40.0 kg/m2.
* Informed consent signed.

Group III:

* Polycystic ovary syndrome phenotype IV (NIH-2012) (http://prevention.nih.gov/workshops/2012/resources.aspx).
* Body mass index between 18.5 and 40.0 kg/m2.
* Informed consent signed.

Group IV:

* Body mass index between 18.5 and 25.0 kg/m2.
* Regular menses.
* Normal gonadotropins and estradiol levels at follicular phase.
* Moderate-vigorous intensity physical activity (> 5 hours per week) with normal energy availability (> 30 kcal/per kg of lean mass).
* Informed consent signed.

Group V:

* No signs or symptoms of hyperandrogenism.
* No exercise or mild intensity physical activity.
* Regular menses.
* Body mass index between 18.5 and 40.0 kg/m2.
* Informed consent signed.

Exclusion Criteria (Groups I-V)

* Oral drugs interfering with ovulation (glucocorticoids, antipsychotics, antidepressants, contraceptives, sex steroids and/or opioids) for the previous 6 months to study inclusion.
* Current pregnancy or lactation, or during the previous 6 months to study inclusion.
* Asherman's syndrome or outflow tract disorders.
* Current smoking or alcohol intake > 40 g per day.
* Previous diagnosis of glucose intolerance, hypertension, dyslipidemia, known heart or lung diseases, kidney disease, liver disease, celiac disease or any other malabsorptive condition, chronic inflammatory disease or malignancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with exercise-associated functional amenorrhea and polycystic ovary syndrome will be consecutively recruited from our Reproductive Endocrinolgy clinic. Those premenopausal adult women are referred to clinic because of symptoms of functional androgen excess such as hirsutism or menstrual dysfunction.
  The control group (Groups IV and V) will include healthy female volunteers recruited - contemporarily with the recruitment of patients - from the hospital's staff and overweight or obese women seeking medical attention in our department.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adipokine and myokine signaling identification | Up to 5 years

SECONDARY OUTCOMES:
Circulating adipokine profile | Up to 5 years
  At fasting and after an oral glucose challenge: Circulating concentrations of Leptin, Adiponectin, Chemerin, Lipocalin-2, Adipsin, Plasminogen Activator Inhibitor (PAI)-1, Monocyte Chemoattractant Protein (MCP)-1, and Soluble Leptin Receptor by multianalyte profiling on the Luminex Magpix system (Luminex Technologies, Austin, USA.).
Appetite regulation hormonal profile | Up to 5 years
  At fasting and after an oral glucose challenge: Circulating concentrations of Amylin, C-Peptide, Ghrelin, Gastric Inhibitory Peptide (GIP), Glucagon-Like Peptide (GLP)-1, Glucagon, IL-6, Insulin, Pancreatic Polypeptide (PP), Peptide YY, Tumor Necrosis Factor (TNF)-α by multianalyte profiling on the Luminex Magpix system (Luminex Technologies, Austin, USA.).
Association between body mass index and sex steroids | Up to 5 years
  Body mass index in in kg/m^2. Sex steroids (including circulating total testosterone, estradiol, androstenedione, dehydroepiandrosterone-sulphate and estrone) measured by liquid chromatography tandem mass spectrometry (LC-MS/MS). Free testosterone will be calculated from total testosterone and sex hormone binding globulin levels.
Association between percentage of fat mass with respect to total body weight and sex steroids | Up to 5 years
  Fat mass% by bioelectric impedanciometry and DEXA. Sex steroids (including circulating total testosterone, estradiol, androstenedione, dehydroepiandrosterone-sulphate and estrone) measured by liquid chromatography tandem mass spectrometry (LC-MS/MS). Free testosterone will be calculated from total testosterone and sex hormone binding globulin levels.
Association between percentage of lean mass with respect to total body weight and sex steroids | Up to 5 years
  Lean mass% by bioelectric impedanciometry and DEXA. Sex steroids (including circulating total testosterone, estradiol, androstenedione, dehydroepiandrosterone-sulphate and estrone) measured by liquid chromatography tandem mass spectrometry (LC-MS/MS). Free testosterone will be calculated from total testosterone and sex hormone binding globulin levels.
Association between body fat depots and sex steroids | Up to 5 years
  Adipose tissue depots will be estimated using a Toshiba Nemio XG SSA-580A Diagnostic Ultrasound System. Minimum sc and preperitoneal fat thicknesses will be measured at the level of the xyphoid process. Maximum sc fat thickness will be measured at the level of the umbilicus. Intraperitoneal fat thickness will be measured placing a probe transversally in the midline of abdomen, 2 cm above the umbilicus. Three measures of ip fat thickness will be obtained: the distance from the fascia of rectus abdominis muscle to the vertebral column, the distance from the peritoneum to the vertebral column, and the distance from the linea alba to the vertebral column. Perirenal fat thickness will be estimated as the distance from the perirenal fascia to the renal surface. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and insulin resistance. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Fasting glucose and insulin levels will be used for calculating the homeostasis model assessment of insulin resistance (HOMA-IR), and the composite insulin sensitivity index will be estimated from the glucose and insulin concentrations measured during the oral glucose tolerance test. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and lipids. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Circulating HDL-cholesterol and phospholipid levels will be measured by enzymatic methods after precipitation of plasma with phosphotungstic acid and Mg2+. Total cholesterol and triglyceride levels will be determined by enzymatic methods. LDL-cholesterol concentrations will be estimated by Friedewald's equation. Circulating apolipoprotein (Apo) AI, Apo B100, and lipoprotein (a) levels will be determined by kinetic immunonephelometry. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and office blood pressure. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Office blood pressure will be determined as the mean of three manual sphygmomanometer readings in the sitting position. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and ambulatory blood pressure monitoring parameters. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Twenty-four-hour ambulatory blood pressure monitoring will be performed using an A&D TM2430EX oscillometric device (A&D Co., Ltd., Tokyo, Japan). The cuff (12 × 22 cm for lean participants, 14 × 30 cm for overweight or obese participants) will placed on the nondominant arm in every woman. The period from 0700 to 2300 h will be considered daytime, and from 2300 until 0700 h the next day will be considered nighttime, reflecting the usual sleeping habits of Spaniards. Systolic, diastolic, and mean blood pressure as well as heart rate will be measured every 20 min during daytime and every 30 min during nighttime. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and cardiovascular autonomic function tests. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Cardiovascular autonomic function will be assessed by the blood pressure and heart rate responses to active standing, and Ewing and Clarke's tests. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and carotid intima-media thickness. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Imaging will be conducted using a high-resolution 7.5-MHz phased-array transducer by the same trained operator in all the participants. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and oxidative stress. | Up to 5 years
  Fat mass, lean mass and body fat depots will be measured as previously described. Oxidative stress profile will be measured by enzymatic assays: Plasma thiobarbituric acid reactive substances, total antioxidant capacity, nitrotyrosine, protein carbonyl groups and erythrocyte glutathione peroxidase levels. Sex steroids will be measured as previously described.
Association between body composition, sex steroids, and microbiome | Up to 5 years
  Participants will be instructed to collect fecal and salivary samples. DNA samples wil be used for massive sequencing of 16S ribosomal DNA (rDNA) amplicons in a MiSeq platform (Illumina). The bacterial diversity will be estimated by using Shannon, Chao 1, Jaccard, and Sorensen indexes with their SDs. Taxonomic affiliations will be assigned by using the RDP_classifier from the Ribosomal Database Project (RDP), and readings with RDP score value <0.8 will be assigned to the upper taxonomic rank, leaving the last rank as unidentified. Sex steroids will be measured as previously described.

CONTACTS AND LOCATIONS:
Overall Officials: Héctor F Escobar-Morreale, PhD, MD, Principal Investigator — Diabetes, Obesity and Human Reproduction Research Group (CIBERDEM), Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS), Madrid, Spain; Manuel Luque-Ramírez, PhD, MD, Principal Investigator — Diabetes, Obesity and Human Reproduction Research Group (CIBERDEM), Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS), Madrid, Spain
Locations (1):
- Endocrinology and Nutrition, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The investigators will deposit any datasets and supplemental materials to a generalist repository. The investigators will refer to the deposited material as an item in the bibliography of any manuscript and number the reference appropriately within the text.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the time of the first manuscript submission.
Access Criteria: Public access

REFERENCES:
- [Background] Ortiz-Flores AE, Luque-Ramirez M, Fernandez-Duran E, Alvarez-Blasco F, Escobar-Morreale HF. Diagnosis of disorders of glucose tolerance in women with polycystic ovary syndrome (PCOS) at a tertiary care center: fasting plasma glucose or oral glucose tolerance test? Metabolism. 2019 Apr;93:86-92. doi: 10.1016/j.metabol.2019.01.015. Epub 2019 Jan 30. PMID 30710572
- [Background] Luque-Ramirez M, Jimenez-Mendiguchia L, Garcia-Cano A, Fernandez-Duran E, de Dios Rosa V, Nattero-Chavez L, Ortiz-Flores AE, Escobar-Morreale HF. Certified testosterone immunoassays for hyperandrogenaemia. Eur J Clin Invest. 2018 Dec;48(12):e13029. doi: 10.1111/eci.13029. Epub 2018 Oct 8. PMID 30229887
- [Background] Insenser M, Murri M, Del Campo R, Martinez-Garcia MA, Fernandez-Duran E, Escobar-Morreale HF. Gut Microbiota and the Polycystic Ovary Syndrome: Influence of Sex, Sex Hormones, and Obesity. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2552-2562. doi: 10.1210/jc.2017-02799. PMID 29897462
- [Background] Escobar-Morreale HF. Polycystic ovary syndrome: definition, aetiology, diagnosis and treatment. Nat Rev Endocrinol. 2018 May;14(5):270-284. doi: 10.1038/nrendo.2018.24. Epub 2018 Mar 23. PMID 29569621
- [Background] Escobar-Morreale HF. The Role of Androgen Excess in Metabolic Dysfunction in Women : Androgen Excess and Female Metabolic Dysfunction. Adv Exp Med Biol. 2017;1043:597-608. doi: 10.1007/978-3-319-70178-3_26. PMID 29224112
- [Background] Montes-Nieto R, Insenser M, Murri M, Fernandez-Duran E, Ojeda-Ojeda M, Martinez-Garcia MA, Luque-Ramirez M, Escobar-Morreale HF. Plasma thiobarbituric acid reactive substances (TBARS) in young adults: Obesity increases fasting levels only in men whereas glucose ingestion, and not protein or lipid intake, increases postprandial concentrations regardless of sex and obesity. Mol Nutr Food Res. 2017 Nov;61(11). doi: 10.1002/mnfr.201700425. Epub 2017 Aug 29. PMID 28722287
- [Background] Escobar-Morreale HF, Martinez-Garcia MA, Montes-Nieto R, Fernandez-Duran E, Temprano-Carazo S, Luque-Ramirez M. Effects of glucose ingestion on circulating inflammatory mediators: Influence of sex and weight excess. Clin Nutr. 2017 Apr;36(2):522-529. doi: 10.1016/j.clnu.2016.01.015. Epub 2016 Jan 29. PMID 26874912
- [Background] Insenser M, Montes-Nieto R, Martinez-Garcia MA, Escobar-Morreale HF. A nontargeted study of muscle proteome in severely obese women with androgen excess compared with severely obese men and nonhyperandrogenic women. Eur J Endocrinol. 2016 Mar;174(3):389-98. doi: 10.1530/EJE-15-0912. Epub 2015 Dec 15. PMID 26671973
- [Background] Borruel S, Molto JF, Alpanes M, Fernandez-Duran E, Alvarez-Blasco F, Luque-Ramirez M, Escobar-Morreale HF. Surrogate markers of visceral adiposity in young adults: waist circumference and body mass index are more accurate than waist hip ratio, model of adipose distribution and visceral adiposity index. PLoS One. 2014 Dec 5;9(12):e114112. doi: 10.1371/journal.pone.0114112. eCollection 2014. PMID 25479351
- [Background] Luque-Ramirez M, Escobar-Morreale HF. Polycystic ovary syndrome as a paradigm for prehypertension, prediabetes, and preobesity. Curr Hypertens Rep. 2014 Dec;16(12):500. doi: 10.1007/s11906-014-0500-6. PMID 25304109
- [Background] Escobar-Morreale HF, Alvarez-Blasco F, Botella-Carretero JI, Luque-Ramirez M. The striking similarities in the metabolic associations of female androgen excess and male androgen deficiency. Hum Reprod. 2014 Oct 10;29(10):2083-91. doi: 10.1093/humrep/deu198. Epub 2014 Aug 7. PMID 25104855
- [Background] Murri M, Insenser M, Luque M, Tinahones FJ, Escobar-Morreale HF. Proteomic analysis of adipose tissue: informing diabetes research. Expert Rev Proteomics. 2014 Aug;11(4):491-502. doi: 10.1586/14789450.2014.903158. Epub 2014 Mar 31. PMID 24684164
- [Background] Murri M, Insenser M, Escobar-Morreale HF. Metabolomics in polycystic ovary syndrome. Clin Chim Acta. 2014 Feb 15;429:181-8. doi: 10.1016/j.cca.2013.12.018. Epub 2013 Dec 22. PMID 24368231
- [Background] Luque-Ramirez M, Marti D, Fernandez-Duran E, Alpanes M, Alvarez-Blasco F, Escobar-Morreale HF. Office blood pressure, ambulatory blood pressure monitoring, and echocardiographic abnormalities in women with polycystic ovary syndrome: role of obesity and androgen excess. Hypertension. 2014 Mar;63(3):624-9. doi: 10.1161/HYPERTENSIONAHA.113.02468. Epub 2013 Dec 9. PMID 24324038
- [Background] Escobar-Morreale HF. Reproductive endocrinology: Menstrual dysfunction--a proxy for insulin resistance in PCOS? Nat Rev Endocrinol. 2014 Jan;10(1):10-1. doi: 10.1038/nrendo.2013.232. Epub 2013 Nov 26. No abstract available. PMID 24275746
- [Background] Insenser M, Escobar-Morreale HF. Proteomics and polycystic ovary syndrome. Expert Rev Proteomics. 2013 Oct;10(5):435-47. doi: 10.1586/14789450.2013.837665. Epub 2013 Oct 3. PMID 24087928
- [Background] Murri M, Insenser M, Bernal-Lopez MR, Perez-Martinez P, Escobar-Morreale HF, Tinahones FJ. Proteomic analysis of visceral adipose tissue in pre-obese patients with type 2 diabetes. Mol Cell Endocrinol. 2013 Aug 25;376(1-2):99-106. doi: 10.1016/j.mce.2013.06.010. Epub 2013 Jun 18. PMID 23791845
- [Background] Luque-Ramirez M, Martinez-Garcia MA, Montes-Nieto R, Fernandez-Duran E, Insenser M, Alpanes M, Escobar-Morreale HF. Sexual dimorphism in adipose tissue function as evidenced by circulating adipokine concentrations in the fasting state and after an oral glucose challenge. Hum Reprod. 2013 Jul;28(7):1908-18. doi: 10.1093/humrep/det097. Epub 2013 Apr 4. PMID 23559188
- [Background] Insenser M, Montes-Nieto R, Murri M, Escobar-Morreale HF. Proteomic and metabolomic approaches to the study of polycystic ovary syndrome. Mol Cell Endocrinol. 2013 May 6;370(1-2):65-77. doi: 10.1016/j.mce.2013.02.009. Epub 2013 Feb 17. PMID 23422073
- [Background] Borruel S, Fernandez-Duran E, Alpanes M, Marti D, Alvarez-Blasco F, Luque-Ramirez M, Escobar-Morreale HF. Global adiposity and thickness of intraperitoneal and mesenteric adipose tissue depots are increased in women with polycystic ovary syndrome (PCOS). J Clin Endocrinol Metab. 2013 Mar;98(3):1254-63. doi: 10.1210/jc.2012-3698. Epub 2013 Feb 5. PMID 23386652
- [Background] Montes-Nieto R, Insenser M, Martinez-Garcia MA, Escobar-Morreale HF. A nontargeted proteomic study of the influence of androgen excess on human visceral and subcutaneous adipose tissue proteomes. J Clin Endocrinol Metab. 2013 Mar;98(3):E576-85. doi: 10.1210/jc.2012-3438. Epub 2013 Jan 24. PMID 23348399
- [Background] Alvarez-Blasco F, Luque-Ramirez M, Escobar-Morreale HF. Diet composition and physical activity in overweight and obese premenopausal women with or without polycystic ovary syndrome. Gynecol Endocrinol. 2011 Dec;27(12):978-81. doi: 10.3109/09513590.2011.579658. Epub 2011 May 24. PMID 21609197
- [Background] Insenser M, Escobar-Morreale HF. Application of proteomics to the study of polycystic ovary syndrome. J Endocrinol Invest. 2011 Dec;34(11):869-75. doi: 10.3275/8108. Epub 2011 Nov 21. PMID 22104628
- [Background] Escobar-Morreale HF, Samino S, Insenser M, Vinaixa M, Luque-Ramirez M, Lasuncion MA, Correig X. Metabolic heterogeneity in polycystic ovary syndrome is determined by obesity: plasma metabolomic approach using GC-MS. Clin Chem. 2012 Jun;58(6):999-1009. doi: 10.1373/clinchem.2011.176396. Epub 2012 Mar 16. PMID 22427353
- [Background] Insenser M, Montes-Nieto R, Vilarrasa N, Lecube A, Simo R, Vendrell J, Escobar-Morreale HF. A nontargeted proteomic approach to the study of visceral and subcutaneous adipose tissue in human obesity. Mol Cell Endocrinol. 2012 Nov 5;363(1-2):10-9. doi: 10.1016/j.mce.2012.07.001. Epub 2012 Jul 14. PMID 22796336
- [Background] Murri M, Luque-Ramirez M, Insenser M, Ojeda-Ojeda M, Escobar-Morreale HF. Circulating markers of oxidative stress and polycystic ovary syndrome (PCOS): a systematic review and meta-analysis. Hum Reprod Update. 2013 May-Jun;19(3):268-88. doi: 10.1093/humupd/dms059. Epub 2013 Jan 9. PMID 23303572
- [Background] Martinez-Garcia MA, Montes-Nieto R, Fernandez-Duran E, Insenser M, Luque-Ramirez M, Escobar-Morreale HF. Evidence for masculinization of adipokine gene expression in visceral and subcutaneous adipose tissue of obese women with polycystic ovary syndrome (PCOS). J Clin Endocrinol Metab. 2013 Feb;98(2):E388-96. doi: 10.1210/jc.2012-3414. Epub 2013 Jan 21. PMID 23337724